CLINICAL TRIAL: NCT00858988
Title: A Randomized, Double-blind, Placebo-controlled Trial of Rifaximin, a Non-absorbable Antibiotic, in the Treatment of Tropical Enteropathy
Brief Title: Trial of Rifaximin in the Treatment of Tropical Enteropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Baylor College of Medicine (Other); Kamuzu University of Health Sciences (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MJM-rifaximin
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Tropical Enteropathy
MeSH Terms: conditions — Sprue, Tropical | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin (Experimental)
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — 100mg of rifaxin for 7 consecutive days, twice daily
  Arms: Rifaximin
Drug: Placebo — twice daily for 7 consecutive days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether rifaximin is effective in the treatment of tropical enteropathy in a population of African children at high risk for this disease.

ELIGIBILITY:
Inclusion Criteria:

* live in single village

Exclusion Criteria:

* acutely malnourished
* acutely ill
* chronic disease

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, Principal Investigator — Washington University School of Medicine
Locations (1):
- Limela, Malawi

RESULTS

PARTICIPANT FLOW:
Groups:
- Rifaximin: Allocated to rifaximin
- Placebo: Allocated to placebo
Period: Randomized and Allocation
Arm/Group | Rifaximin | Placebo
Started | 74 | 73
Completed | 74 | 73
Not Completed | 0 | 0
Period: Analysis
Arm/Group | Rifaximin | Placebo
Started | 74 | 73
Completed | 72 | 72
Not Completed | 2 | 1
Not completed — Lactulose unable to be detected in urine | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifaximin | Placebo | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Customized [Mean (Standard Deviation); unit: Months]
  Age | 47.6 (6.5) | 46.8 (7.6) | 47.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 40 | 43 | 83

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Urinary L:M Ratio Before and After the Intervention
Description: To initiate the test, each child drank a 100 ml sugar solution containing 5 g lactulose, 1 g mannitol, 1 g sucralose, and 10 g sucrose. Children remained at the village research site for 4 h after ingestion of the sugar solution, during which time all of the child's urine was collected in a sterile cup with 10 mg merthiolate added to limit the bacterial degradation of excreted sugars. The reported values for normal L:M range from 0.03 to 0.12. A value of ≥0.10 was chosen to be indicative of tropical enteropathy. This test was performed at enrollment and then 28 days later.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Ratio of lactulose-to-mannitol (L:M) exc
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 72 | 72
Ratio of lactulose-to-mannitol (L:M) exc | -0.01 (0.12) | 0.02 (0.16)

ADVERSE EVENTS:
Arm/Group | Rifaximin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes